CLINICAL TRIAL: NCT02700620
Title: Individually Tailored Web-based Cbt for Eating Disorders and the Role of Knowledge Acquisition
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Linkoeping University (Other Government)
Responsible Party: Principal Investigator, Gerhard Andersson, Professor, Linkoeping University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2014-426-31
Record Dates: First submitted 2015-10-26; First posted 2016-03-07 (Estimated); Last update posted 2023-12-14 (Actual); Status verified 2023-12

CONDITIONS: Eating Disorders; Bulimia
Keywords: emotional eating; restrictive eating; body dissatisfaction
MeSH Terms: conditions — Feeding and Eating Disorders; Bulimia; Emotional Eating

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment group (Experimental): Internet-delivered CBT
  Interventions: Behavioral: Internet-delivered CBT
- Control group (No Intervention): Waitlist control

INTERVENTIONS:
Behavioral: Internet-delivered CBT — Guided internet treatment
  Arms: Treatment group

SUMMARY:
Background: Previous studies on Internet-based treatment with eating disorders have shown promising results.

Objective: The first aim of this study was to investigate the effects of a tailored therapist guided internet-based treatment for individuals with eating disorders. The second aim was to examine the role of knowledge acquisition.

Method: 138 participants were recruited. Screening consisted of online questionnaires followed by a telephone interview. A total of 92 participants were included after a semi-structured diagnostic interview and randomized to an 8 week treatment program (n=46) or to a control condition (n=46). Treatment consisted of individually prescribed cognitive behaviour therapy text modules in conjunction with online therapist guidance. The control group consisted of a waitlist who later received treatment.

DETAILED DESCRIPTION:
As above

ELIGIBILITY:
Inclusion Criteria:

* Have reoccurring eating disorder uns or bulimia
* BMI above 17,5

Exclusion Criteria:

* Suicide prone
* Ongoing psychological treatment

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2015-01; Primary Completion 2017-06 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Eating Disorders Examination Questionnaire | post (8 weeks)

SECONDARY OUTCOMES:
Quality of Life Inventory (QOLI) | Pre and post (8 weeks)
Body Shape Questionnaire (BSQ) | post (8 weeks)
Patient Health Questionnaire (PHQ-9) | post (8 weeks)
Generalised Axiety Disorder Assessment (GAD-7) | post (8 weeks)
Satisfaction With Life Scales (SWLS) | post (8 weeks)
Expectancy/Credibility Questionnaire (CEQ) | post (8 weeks)

IPD SHARING:
Plan to Share IPD: Yes
Primary outcomes and background info on request.

REFERENCES:
- [Derived] Strandskov SW, Ghaderi A, Andersson H, Parmskog N, Hjort E, Warn AS, Jannert M, Andersson G. Effects of Tailored and ACT-Influenced Internet-Based CBT for Eating Disorders and the Relation Between Knowledge Acquisition and Outcome: A Randomized Controlled Trial. Behav Ther. 2017 Sep;48(5):624-637. doi: 10.1016/j.beth.2017.02.002. Epub 2017 Mar 2. PMID 28711113